CLINICAL TRIAL: NCT04019210
Title: Modified Trabeculectomy a New Procedure for Glaucoma Surgery
Brief Title: Modified Trabeculectomy for Glaucoma Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hassan Lotfy Fahmy, Clinical Professor, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2323298
Record Dates: First submitted 2019-07-07; First posted 2019-07-15 (Actual); Last update posted 2019-07-15 (Actual); Status verified 2019-07

CONDITIONS: IOP Decreased
MeSH Terms: conditions — Ocular Hypotension

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MODIFIED TRABECULECTOMY (Experimental): Recta-angular scleral flap (one half the scleral thickness) is dissected,reaching 2 mm into the cornea. The dissection through the cornea is carried out with great care, leaving only thin corneal stroma over Descement's membrane.
  Application of direct heat cautery using a prob Imm in size (the prob was heated for 45 seconds) the cautery was applied at 4 points two of them just in front of blue corneal line and the other two at 2 mm anterior to the blue line, the diameter of each point is 1 - 1.5 mm.
  Interventions: Procedure: MODIFIED TRABECULECTOMY

INTERVENTIONS:
Procedure: MODIFIED TRABECULECTOMY — Rectangular scleral flap

SUMMARY:
A combination of hypotony, flat anterior chamber and choroidal detachment is the most common complications after filtering surgery. The purpose of this study is to present a new modification in standard trabeculectomy technique to reduce such complications.

DETAILED DESCRIPTION:
Recta-angular scleral flap (one half the scleral thickness) is dissected,reaching 2 mm into the cornea. The dissection through the cornea is carried out with great care, leaving only thin corneal stroma over Descement's membrane.

Application of direct heat cautery using a prob Imm in size (the prob was heated for 45 seconds) the cautery was applied at 4 points two of them just in front of blue corneal line and the other two at 2 mm anterior to the blue line, the diameter of each point is 1 - 1.5 mm. The horizontal distance between each point is 3.5 mm Figure(1). The application of the cautery continue till the color of the tissue becomes brown.

Then with aid of a 23-gauge needle we penetrate these cauterized points to create 4 holes, each of them is nearly 0.3-0.5 mm in length (the opening of each hole takes the shape of a slit). Through one of these holes iridectomy is done.

These holes drain the aqueous under the scleral flap with anatomical preservation of tissue in between.

Close the scleral flap by two 10-0 nylon suture.

ELIGIBILITY:
Inclusion Criteria:

* 1ery glacouma

Exclusion Criteria:

* Previous surgery

Ages: 30 Years to 62 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 17 (Estimated)
Dates: Start 2015-10 (Actual); Primary Completion 2019-11 (Estimated); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
IOP | 6 month
  Decreased IOP with normal depth anterior chamber measured by Tonopen

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut U, Asyut, Egypt